CLINICAL TRIAL: NCT03739203
Title: A Double-Blind, Placebo-Controlled Study of Cariprazine as an Adjunct to Antidepressants in the Treatment of Patients With Major Depressive Disorder Who Have Had an Inadequate Response to Antidepressants Alone
Brief Title: The Objective of This Study is to Evaluate the Efficacy, Safety and Tolerability of Cariprazine as an Adjunctive Treatment to Antidepressant Therapy (ADT) in Patients With Major Depressive Disorder (MDD) Who Have Had an Inadequate Response to Antidepressants Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3111-302-001; 2018-003164-31 (EudraCT Number)
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Major Depressive Disorder
Keywords: MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo + ADT (Placebo Comparator): Cariprazine matching placebo capsules, orally, once daily in addition to their ongoing antidepressant therapy (ADT) [same antidepressant and dose of ADT they were on at the Baseline] during the Double-blind Treatment Period, up to Week 6.
  Interventions: Drug: Placebo; Drug: Antidepressant Therapy (ADT)
- Cariprazine 1.5 mg/day + ADT (Experimental): Cariprazine 1.5 mg capsules, orally, once daily in addition to their ongoing ADT (same antidepressant and dose of ADT they were on at the Baseline) during the Double-blind Treatment Period, up to Week 6.
  Interventions: Drug: Cariprazine; Drug: Antidepressant Therapy (ADT)
- Cariprazine 3 mg/day + ADT (Experimental): Cariprazine 1.5 mg capsules, orally, once daily for 2 weeks starting at the Baseline, titrated to 3.0 mg capsules, orally, once daily from Week 2 through Week 6 in addition to their ongoing ADT (same antidepressant and dose of ADT) during the Double-blind Treatment Period, up to Week 6.
  Interventions: Drug: Cariprazine; Drug: Antidepressant Therapy (ADT)

INTERVENTIONS:
Drug: Cariprazine — Cariprazine supplied in capsules
  Other Names: VRAYLAR®
  Arms: Cariprazine 1.5 mg/day + ADT; Cariprazine 3 mg/day + ADT
Drug: Placebo — Placebo supplied in capsules
  Arms: Placebo + ADT
Drug: Antidepressant Therapy (ADT) — ADT as prescribed by the physician per standard of care in clinical practice.

SUMMARY:
The objective of this study is to evaluate the efficacy, safety and tolerability of cariprazine as an adjunctive treatment to antidepressant therapy (ADT) in patients with MDD who have had an inadequate response to antidepressants alone.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained.
* Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable (eg, Written Authorization for Use and Release of Health and Research Study Information [US sites] and written Data Protection consent [EU sites]).
* Participant must be an outpatient at the time of Visit 1 (Screening).
* Participant meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD based on Structured Clinical Interview for DSM-5 (SCID-5), with a current major depressive episode of at least 8 weeks and not exceeding 24 months in duration at Visit 1/Screening. A diagnosis of MDD with psychotic features will be acceptable.
* Diagnosis of MDD confirmed through a formal adjudication process.
* Participant demonstrates ability to follow study instructions and likely to complete all required visits.
* Participant must have an inadequate response, as measured by the modified antidepressant treatment response questionnaire (ATRQ), to 1 to 3 antidepressants administered during the current episode at an adequate dose (as per package insert) and for at least 6 weeks duration, with at least one dose escalation during the current depressive episode.
* Only one antidepressant (of sufficient dose per package insert and taken for at least 6 weeks) will be allowed at randomization and Participants must agree to continue taking the same ADT dosing regimen through completion of Visit 6/early termination (ET). Participants who are taking more than one antidepressant at Screening, regardless of the indication, will need to discontinue all other antidepressants prior to Visit 2 (Baseline).
* Male and female Participants must agree to use a medically acceptable and highly effective method of birth control during the course of the entire study.
* Women of childbearing potential (only) must have a negative serum β-human chorionic gonadotropin pregnancy test prior to Visit 2.

Exclusion Criteria:

* Diagnosis of any current psychiatric diagnosis other than MDD (including those with current intellectual development disability) with the exception of specific phobias.
* Participant has a history of intolerance or hypersensitivity to cariprazine or other drugs of the same class or to rescue medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 752 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (112):
- United States (58):
  - Harmonex /ID# 236936, Dothan, Alabama
  - Woodland International Research Group /ID# 236349, Little Rock, Arkansas
  - California Pharmaceutical Research Institute /ID# 236731, Anaheim, California
  - Axiom Research /ID# 236267, Colton, California
  - Global Clinical Trials /ID# 235059, Costa Mesa, California
  - Collaborative Neuroscience Research - Orange County /ID# 237637, Garden Grove, California
  - Behavioral Research Specialists, LLC /ID# 236622, Glendale, California
  - Sun Valley Research Center /ID# 236560, Imperial, California
  - North County Clinical Research /ID# 235014, Oceanside, California
  - Excell Research, Inc /ID# 237717, Oceanside, California
  - NRC Research Institute /ID# 234632, Orange, California
  - Anderson Clinical Research /ID# 236624, Redlands, California
  - Syrentis Clinical Research /ID# 237408, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc. /ID# 236636, Sherman Oaks, California
  - Schuster Medical Research Institute /ID# 236445, Sherman Oaks, California
  - Pacific Clinical Research Management Group /ID# 234378, Upland, California
  - MCB Clinical Research Centers /ID# 236927, Colorado Springs, Colorado
  - CT Clinical Research /ID# 234638, Cromwell, Connecticut
  - Innovative Clinical Research /ID# 235186, Fort Lauderdale, Florida
  - Gulfcoast Clinical Research Center /ID# 236280, Fort Myers, Florida
  - Innova Clinical Trials /ID# 237376, Miami, Florida
  - International Research Associates, LLC /ID# 237410, Miami, Florida
  - Medical Research Group of Central Florida /ID# 237326, Orange City, Florida
  - Clinical Neuroscience Solutions, Inc /ID# 236604, Orlando, Florida
  - Space Coast Neuropsychiatric Research Institute /ID# 235766, Palm Bay, Florida
  - Atlanta Center for Medical Research /ID# 234696, Atlanta, Georgia
  - Institute for Advanced Medical Research /ID# 234992, Atlanta, Georgia
  - iResearch Savannah /ID# 236082, Savannah, Georgia
  - Iris Research Inc. /ID# 234995, Smyrna, Georgia
  - AMR Conventions Research /ID# 236262, Naperville, Illinois
  - Collective Medical Research /ID# 236397, Prairie Village, Kansas
  - Boston Clinical Trials /ID# 236558, Boston, Massachusetts
  - BTC of New Bedford /ID# 236381, New Bedford, Massachusetts
  - The Coastal Research Associates Inc /ID# 235056, South Weymouth, Massachusetts
  - Sisu at Renaissance Medical Group /ID# 236198, Springfield, Massachusetts
  - Center for Emotional Fitness /ID# 236630, Cherry Hill, New Jersey
  - Bio Behavioral Health, Inc /ID# 238209, Toms River, New Jersey
  - SPRI Clinical Trails /ID# 236657, Brooklyn, New York
  - Bioscience Research /ID# 234961, Mount Kisco, New York
  - Fieve Clinical Research, Inc. /ID# 236632, New York, New York
  - Eastside Comprehensive Medical Center LLC /ID# 236094, New York, New York
  - Clinical Trials America /ID# 237636, Hickory, North Carolina
  - Quest Therapeutics of Avon Lake /ID# 236281, Avon Lake, Ohio
  - Patient Priority Clinical Sites, LLC /ID# 236743, Cincinnati, Ohio
  - North Star Medical Research LL /ID# 235076, Middleburg Heights, Ohio
  - CincyScience /ID# 236387, West Chester, Ohio
  - Lynn Health Science Institute (LHSI) /ID# 237612, Oklahoma City, Oklahoma
  - Central States Research /ID# 238295, Tulsa, Oklahoma
  - Oregon Ctr for Clin Inv /ID# 237463, Salem, Oregon
  - Keystone Clinical Studies LLC /ID# 238153, Plymouth Meeting, Pennsylvania
  - Psychiatric Consultants PC /ID# 235838, Franklin, Tennessee
  - Research Strategies of Memphis /ID# 236629, Memphis, Tennessee
  - Earle Research /ID# 236660, Friendswood, Texas
  - AIM Trials /ID# 236366, Plano, Texas
  - Clinical Trials of Texas, Inc /ID# 237864, San Antonio, Texas
  - Family Psychiatry of The Woodlands /ID# 236423, The Woodlands, Texas
  - Woodstock Research Center /ID# 236653, Woodstock, Vermont
  - SSM Health Dean Medical Group /ID# 238103, Madison, Wisconsin
- Canada (4):
  - Chatham-Kent Clinical Trials /ID# 235707, Chatham, Ontario
  - Introspect Clinical Research Centre /ID# 235987, Ottawa, Ontario
  - Recherches Neuro-Hippocampe Inc. d/b/a Ottawa Memory Clinic /ID# 235890, Ottawa, Ontario
  - Diex Recherche Sherbrooke Inc. /ID# 234385, Sherbrooke, Quebec
- Czechia (7):
  - Medical Services Prague /ID# 235109, Prague, Praha, Hlavni Mesto
  - Saint Anne s.r.o. /ID# 235060, Brno
  - MUDr. Marta Holanova /ID# 235126, Brno
  - Neuropsychiatriehk s.r.o. /ID# 236195, Hradec Králové
  - A-SHINE s.r.o. /ID# 236370, Pilsen
  - CLINTRIAL s.r.o. /ID# 237794, Prague
  - INEP medical s.r.o. /ID# 236291, Prague
- Finland (6):
  - Helsingin psykiatripalvelu /ID# 235090, Helsinki
  - Mederon Oy /ID# 235057, Helsinki
  - Savon Psykiatripalvelu Oy /ID# 235028, Kuopio
  - Oulu Mentalcare Oy /ID# 235089, Oulu
  - Satakunnan Psykiatripalvelu Oy /ID# 234936, Rauma
  - Psykiatri- ja psykologikeskus Mentoria /ID# 235091, Tampere
- Poland (16):
  - Centrum Medyczne Luxmed /ID# 235110, Lublin, Lublin Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 237466, Gdansk, Pomeranian Voivodeship
  - Zachodniopomorski Instytut Psychoterapii /ID# 236549, Szczecin, West Pomeranian Voivodeship
  - Wlokiennicza Med /ID# 235105, Bia?ystok
  - MlynowaMed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk /ID# 235065, Bialystok
  - Przychodnia Srodmiescie Sp. Z o.o. /ID# 236197, Bydgoszcz
  - Med-Art /Id# 234986, Bydgoszcz
  - Poradnia Zdrowia Psychicznego /ID# 234750, Chełmno
  - Centrum Zdrowia Psychicznego BioMed - Jan Latala /ID# 235064, Kielce
  - Nzop Mentis /Id# 235062, Leszno
  - Centrum Medyczne Neuromedica /ID# 235615, Lublin
  - Krzysztof Klinke Prywatny Gabinet Psychiatryczny /ID# 235061, Sosnowiec
  - Gabinet Lekarski Torunskie Centrum Psychiatrii Neuromed /ID# 235001, Torun
  - Osrodek Badan Klinicznych Clinsante /ID# 234990, Torun
  - Przychodnia Lekarsko-Psychologiczna PERSONA /ID# 235007, Wroclaw
  - Gabinet Lekarski Psychiatryczny Ireneusz Kaczorowski /ID# 234851, Bełchatów, Łódź Voivodeship
- INSPIRA Clinical Research /ID# 234542, San Juan, Puerto Rico
- Serbia (12):
  - Military Medical Academy /ID# 237062, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 237747, Belgrade, Beograd
  - University Clinical Center of Nis /ID# 236973, Niš, Nisavski Okrug
  - University Clinical Center Kragujevac /ID# 237750, Kragujevac, Sumadijski Okrug
  - University Clinical Center Kragujevac /ID# 237752, Kragujevac, Sumadijski Okrug
  - University Clinical Center Kragujevac /ID# 237753, Kragujevac, Sumadijski Okrug
  - Bel Medic - General Hospital /ID# 236171, Belgrade
  - Clinical Hospital Center Dr Dragisa Misovic - Dedinje /ID# 234299, Belgrade
  - Institute of Mental Health /ID# 236481, Belgrade
  - Special Hospital for Psychiatric Diseases Kovin /ID# 234691, Kovin
  - Specialized Hospital for Neuropsychiatric Diseases Sveti Vracevi /ID# 234716, Novi Kneževac
  - Special Psychiatric Hospital /ID# 235152, Vršac
- Slovakia (8):
  - J&J SMART Ltd. /ID# 235902, Bratislava
  - Psychiatrická ambulancia MENTUM /ID# 235020, Bratislava
  - Vavrusova Consulting s.r.o. /ID# 235022, Bratislava
  - EPAMED s.r.o. /ID# 234830, Košice
  - Liptovska nemocnica s poliklinikou MUDr. Ivana Stodolu Liptovsky Mikulas /ID# 235216, Liptovský Mikuláš
  - Psycholine s.r.o /ID# 235081, Rimavská Sobota
  - Centrum zdravia R.B.K sro /ID# 235085, Svidník
  - Crystal Comfort s.r.o. /ID# 235083, Vranov nad Topľou

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Riesenberg R, Yeung PP, Rekeda L, Sachs GS, Kerolous M, Fava M. Cariprazine for the Adjunctive Treatment of Major Depressive Disorder in Patients With Inadequate Response to Antidepressant Therapy: Results of a Randomized, Double-Blind, Placebo-Controlled Study. J Clin Psychiatry. 2023 Aug 16;84(5):22m14643. doi: 10.4088/JCP.22m14643. PMID 37585254
- See also: VRAYLAR® (cariprazine) capsules prescribing information. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 752 participants were enrolled, of which 751 took ≥1 dose of double-blind investigational product and were included in the Safety Population. One participant was randomized but did not receive treatment and was excluded from the study analyses. At the end of treatment in the Double-blind Period, participants continued on their background antidepressant therapy (ADT) and entered the Safety Follow-up Period.
Period: Double-blind Treatment Period (6 Weeks)
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
Started | 250 | 250 | 251
Modified Intent-to Treat (mITT) Population (mITT population included all randomized participants who had ≥1 postbaseline assessment of the Montgomery-Asberg Depression Rating Scale (MADRS) total score.) | 249 | 250 | 251
Completed | 235 | 233 | 226
Not Completed | 15 | 17 | 25
Not completed — Adverse Event | 6 | 9 | 13
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 4 | 6
Not completed — Protocol Deviation | 1 | 0 | 1
Not completed — Non-compliance With Study Drug | 1 | 3 | 1
Not completed — Reason not Specified | 1 | 0 | 1
Period: Safety Follow-Up Period (4 Weeks)
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
Started (As per protocol-defined criteria, some of the participants discontinued from the Double-blind Period but entered the Safety Follow-up Period.) | 242 | 242 | 242
Completed | 240 | 240 | 238
Not Completed | 2 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Death | 1 | 0 | 0
Not completed — Reason not Specified | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants in the randomized population who took ≥1 dose of double-blind investigational product.
Groups:
- Placebo + ADT: Cariprazine matching placebo capsules, orally, once daily in addition to their ongoing ADT (same antidepressant and dose of ADT they were on at the Baseline) during the Double-blind Treatment Period, up to Week 6.
- Total: Total of all reporting groups
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT | Total
Number analyzed (Participants) | 250 | 250 | 251 | 751
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (12.12) | 45.0 (12.95) | 45.8 (12.45) | 45.7 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 185 | 197 | 573
  Male | 59 | 65 | 54 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 38 | 34 | 102
  Not Hispanic or Latino | 220 | 212 | 217 | 649
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 4 | 0 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 29 | 32 | 22 | 83
  White | 217 | 216 | 221 | 654
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Montgomery-Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The MADRS is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants are rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item is scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity. The total score ranges from 0 to 60 with a higher score indicating more depression. Population: mITT Population included all randomized participants who had ≥1 postbaseline assessment of the MADRS total score.
  score on a scale
    number analyzed (Participants) | 249 | 250 | 251 | 750
    (all) | 32.99 (4.789) | 32.00 (4.246) | 32.25 (4.688) | 32.41 (4.593)
Clinical Global Impression-Severity (CGI-S) Scale Score [Mean (Standard Deviation); unit: score on a scale] — The CGI-S is a clinician-rated scale used to rate the severity of the participant's current state of mental illness compared with MDD population. The participant was rated on a scale from 1 to 7, where 1=normal, not at all ill and 7=among the most extremely ill participants. Higher score indicates worsening of mental illness. Population: mITT Population included all randomized participants who had ≥1 postbaseline assessment of the MADRS total score.
  score on a scale
    number analyzed (Participants) | 249 | 250 | 251 | 750
    (all) | 4.67 (0.599) | 4.61 (0.586) | 4.65 (0.654) | 4.64 (0.614)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in the MADRS (Montgomery-Åsberg Depression Rating Scale) Total Score
Description: The MADRS is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants were rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item was scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity. The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change from Baseline indicates improvement. Mixed-effects Model for Repeated Measures (MMRM) was used for analyses.
Time Frame: Baseline and Week 6
Population: mITT Population included all randomized participants who had ≥1 postbaseline assessment of the MADRS total score. Overall number of participants analyzed are the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
Number analyzed (Participants) | 236 | 237 | 231
score on a scale | -13.4 (0.70) | -13.8 (0.69) | -14.8 (0.70)
Statistical Analysis 1: Comparison: Placebo + ADT vs Cariprazine 1.5 mg/Day + ADT; Test type: Superiority; p = 0.6798, MMRM — p-value estimated by Mixed-effects Model for Repeated Measure from test of no difference between cariprazine dose group and placebo at Week 6; MMRM=Fixed effects:treatment group(TG),ADT failure category,visit,TG-by-visit;Covariates:Baseline(BL)value& BL by-visit interaction; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-2.10 to 1.37], Standard Error of Mean 0.88
Statistical Analysis 2: Comparison: Placebo + ADT vs Cariprazine 3 mg/Day + ADT; Test type: Superiority; p = 0.1245, MMRM — [p-value comment as in outcome 1, analysis 1]; MMRM=Fixed effects:treatment group(TG), ADT failure category,visit,TG-by-visit;Covariates:Baseline(BL)value& BL by-visit interaction; Least Squares Mean Difference = -1.4, 95% CI 2-sided [-3.11 to 0.38], Standard Error of Mean 0.89

2. Secondary Outcome: Change From Baseline to Week 6 in the Clinical Global Impressions-Severity (CGI-S) Score
Description: The CGI-S is a clinician-rated scale used to rate the severity of the participant's current state of mental illness compared with MDD population. The participant was rated on a scale from 1 to 7, where 1=normal, not at all ill and 7=among the most extremely ill participants. Higher score indicates worsening of mental illness. A negative change from Baseline indicates improvement. MMRM was used for analyses.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
Number analyzed (Participants) | 236 | 237 | 231
score on a scale | -1.4 (0.09) | -1.4 (0.09) | -1.6 (0.09)
Statistical Analysis 1: Comparison: Placebo + ADT vs Cariprazine 1.5 mg/Day + ADT; Test type: Superiority; p = 0.5152, MMRM — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.29 to 0.15], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo + ADT vs Cariprazine 3 mg/Day + ADT; Test type: Superiority; p = 0.0573, MMRM — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 2]; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.43 to 0.01], Standard Error of Mean 0.11

ADVERSE EVENTS:
Time Frame: First dose of study drug until 30 days after the last dose of study drug (up to 12 weeks)
Description: Safety Population included all participants in the randomized population who took ≥1 dose of double-blind investigational product.
Arm/Group | Placebo + ADT | Cariprazine 1.5 mg/Day + ADT | Cariprazine 3 mg/Day + ADT
All-Cause Mortality (participants affected / at risk) | 1/250 | 0/250 | 0/251
Serious Adverse Events (participants affected / at risk) | 2/250 | 3/250 | 1/251
Other Adverse Events (participants affected / at risk) | 54/250 | 70/250 | 85/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + ADT (N=250) | Cariprazine 1.5 mg/Day + ADT (N=250) | Cariprazine 3 mg/Day + ADT (N=251)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + ADT (N=250) | Cariprazine 1.5 mg/Day + ADT (N=250) | Cariprazine 3 mg/Day + ADT (N=251)
NAUSEA (Gastrointestinal disorders) | 10 (15) | 14 (16) | 16 (21)
AKATHISIA (Nervous system disorders) | 9 (10) | 19 (19) | 29 (34)
HEADACHE (Nervous system disorders) | 27 (33) | 24 (32) | 27 (40)
SOMNOLENCE (Nervous system disorders) | 11 (11) | 12 (13) | 17 (17)
INSOMNIA (Psychiatric disorders) | 9 (12) | 16 (18) | 25 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT03739203/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03739203/SAP_001.pdf